CLINICAL TRIAL: NCT02791503
Title: CROSSFIRE Trial: Crossatlantic Randomized Controlled Trial Comparing Outcome in Survival After Systemic Plus Focal Therapy for Inoperable Pancreatic Carcinoma: Radiotherapy Versus Irreversible Electroporation
Brief Title: CROSSFIRE Trial: Comparing the Efficacy of Irreversible Electroporation With Radiotherapy
Acronym: CROSSFIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. M.R. Meijerink (Other)
Responsible Party: Sponsor-Investigator, Dr. M.R. Meijerink, dr., Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL55158.029.15
Record Dates: First submitted 2016-05-17; First posted 2016-06-06 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Neoplasm
Keywords: Irreversible electroporation (IRE; Stereotactic ablative radiotherapy (SABR; Efficacy; Tumor ablation; Chemotherapy; Locally advanced pancreatic cancer (LAPC)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IRE group (Experimental): FOLFIRINOX + IRE For patients diagnosed with LAPC, a combination of chemotherapy plus local tumor destruction using irreversible electroporation (IRE), a novel tumor ablation technique, has recently shown great promise. IRE is based on permeabilization of the cell membrane through electrical pulses leading to apoptosis. Theoretically, IRE only affects viable tumor tissue, leaving surrounding vital structures relatively intact. It is therefore considered to cause less morbidity than thermal ablative strategies.
  Interventions: Procedure: Irreversible electroporation (IRE)
- SABR group (Active Comparator): FOLFIRINOX + SABR Focal therapy using external beam radiation therapy (EBRT) may further improve survival, but outcome remains poor. Stereotactic ablative radiotherapy (SABR) is a form of EBRT that has important advantages over conventional radiotherapy such as a more precise and greater biological dose delivery and hence less toxicity and presumably better outcome.
  Interventions: Procedure: Stereotactic ablative radiotherapy (SABR)

INTERVENTIONS:
Procedure: Irreversible electroporation (IRE) — IRE is based on permeabilization of the cell membrane through electrical pulses leading to apoptosis. Theoretically, IRE only affects viable tumor tissue, leaving surrounding vital structures relatively intact. It is therefore considered to cause less morbidity than thermal ablative strategies.
  Other Names: NanoKnife
  Arms: IRE group
Procedure: Stereotactic ablative radiotherapy (SABR) — Stereotactic ablative radiotherapy (SABR) is a form of external beam radiation that has important advantages over conventional radiotherapy such as a more precise and greater biological dose delivery and hence less toxicity and presumably better outcome.
  Arms: SABR group

SUMMARY:
Irreversible electroporation (IRE) is a promising new ablation technique to fight pancreatic cancer. The primary aim of the CROSSFIRE trial is to compare the efficacy (in terms of overall survival) of FOLFIRINOX and IRE (experimental arm) to the efficacy of FOLFIRINOX and stereotactic ablative radiotherapy (SABR) (control arm) in patients with locally advanced, non-resectable, non-metastasized, pancreatic cancer (LAPC). Secondary outcomes are progression free survival, safety/toxicity, immunomodulation, tumor marker Cancer Antigen (CA) 19.9, quality of life (QoL), and total direct and indirect costs for each treatment arm (cost-effectiveness analysis).

DETAILED DESCRIPTION:
Pancreatic cancer has the highest mortality rate of all major cancers; 94% of pancreatic cancer patients will die within five years of diagnosis, 74% within the first year of diagnosis; only 6% will survive for more than five years. Surgical resection is the only curative option. However, about 40% present with non-metastatic locally advanced pancreatic carcinoma (LAPC; AJCC stage III). These patients are not eligible for surgical resection because the tumor involves major blood vessels such as the superior mesenteric artery, celiac axis, common hepatic artery and/or portal vein. These patients are currently treated with palliative chemotherapy as first line therapy. Focal therapy using external beam radiation therapy (EBRT) may further improve survival, but outcome remains poor. Stereotactic ablative radiotherapy (SABR) is a form of EBRT that has important advantages over conventional radiotherapy such as a more precise and greater biological dose delivery and hence less toxicity and presumably better outcome.

For patients diagnosed with LAPC, a combination of chemotherapy plus local tumor destruction using irreversible electroporation (IRE), a novel tumor ablation technique, has recently shown great promise. IRE is based on permeabilization of the cell membrane through electrical pulses leading to apoptosis. Theoretically, IRE only affects viable tumor tissue, leaving surrounding vital structures relatively intact. It is therefore considered to cause less morbidity than thermal ablative strategies.

The CROSSFIRE-trial is a prospective, randomized controlled phase-II/III trial.The primary aim of this study is to compare the efficacy of chemotherapy and IRE (experimental arm) to the efficacy of chemotherapy and radiation (control arm) in patients with locally advanced, non-resectable, non-metastasized, pancreatic cancer.

In total, 138 patients with histologically proven locally advanced pancreatic adenocarcinoma (AJCC stage III), aged ≥ 18 years will be included. Patients with a specific cardiac history (arrhythmias, pacemaker), pre-existent ECG-abnormalities and/or non-retrievable metallic self-expanding biliary stents are excluded from participation. Patients will be randomly allocated to receive either chemotherapy and radiation (control arm) or chemotherapy and IRE (experimental arm).

ELIGIBILITY:
Inclusion Criteria:

* Radiologic confirmation of LAPC by at least ceCT of chest and abdomen (with the upper abdomen scanned according to a dedicated 3mm slice multiphase pancreatic tumor protocol);
* Maximum tumor diameter ≤ 5 cm;
* Histological or cytological confirmation of pancreatic adenocarcinoma;
* Age > 18 years;
* ASA-classification 0 - 3; World Health Organisation scale (WHO) performance status 0 - 1 ;
* Adequate bile drainage in case of biliary obstruction;
* Written informed consent;

Exclusion Criteria:

* Resectable pancreatic adenocarcinoma as discussed by our multidisciplinary hepatobiliary team;
* The presence of suspect lymph nodes
* Stage IV pancreatic carcinoma;
* Trans-mucosal tumor invasion into surrounding duodenum or stomach;
* History of epilepsy;
* History of cardiac disease:

  * Congestive heart failure >NYHA class 2;
  * Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening);
  * Ventricular cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers for antihypertensive regimen are permitted; atrial fibrillation is not contra-indicated);
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen;
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites);
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0);
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment;
* Immunotherapy prior to the procedure;
* Radiotherapy prior to study enrollment;
* Previous surgical therapy for pancreatic cancer;
* Second primary malignancy, except adequately treated non-melanoma skin cancer, in situ carcinoma of the cervis uteri or other malignancies treated at least 5 years previously without signs of recurrence;
* Allergic to contrast agent.
* Any implanted stimulation device;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study;
* Non-removable Self Expanding Metal biliary Stent (SEMS), which cannot be removed during surgery.
* Contra-indications for MRI since no safety data for 0.35 Tesla MRI scanners are available on electronic devices such as pacemakers or implanted defibrillators, deep brain stimulators, cochlear implants, this constitutes an absolute contraindication for this study, even for devices that have been considered safe for MRI scans with higher field strengths.

  * Patients who have a metallic foreign body in their eye, or who have an aneurysm clip in their brain, cannot have an MRI scan since the magnetic field may dislodge the metal
  * Patients with severe claustrophobia may not be able to tolerate an MRI scan
  * Patients with a hip prosthesis will not be eligible for the MRI scan

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-05-30; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of date of death from any cause, assessed up to 100 months

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Untreatable progression-free survival (uPFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] within 90 days after the procedure (IRE/SABR)
Pain assessment | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months by using the a scale
  Pain assessment by using a scale.
Cost-effectiveness analysis | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Direct and indirect total cost of care for both treatment arms (cost-effectiveness analysis);
Quality of life of patients treated with IRE/SABR | From date of randomization until the date of date of death from any cause, whichever came first, assessed up to 100 months by using questionnaires
  Assessing quality of life by using questionnaires.
Change in immune status and reactivity after the procedure (IRE/SABR) by assessing the level of immune cells pre- and post-IRE | Up to 3 months post-procedure
  Measurement of circulating immune cells pre- and post-IRE
Tumor marker CA 19.9 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bart Geboers, Amsterdam, Non-US/Non-Canadian, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Geboers B, Timmer F, Vos D, Scheffer H, Bakker J, Ruarus A, Vroomen L, Stam A, Lougheed S, Schouten E, Puijk R, van den Tol P, Lagerwaard F, de Vries J, Bruynzeel A, Meijerink M, de Gruijl T. Systemic immunomodulation by irreversible electroporation versus stereotactic ablative body radiotherapy in locally advanced pancreatic cancer: the CROSSFIRE trial. J Immunother Cancer. 2025 Mar 26;13(3):e010222. doi: 10.1136/jitc-2024-010222. PMID 40139834
- [Derived] Timmer FEF, Geboers B, Ruarus AH, Vroomen LGPH, Schouten EAC, van der Lei S, Vos DJW, Dijkstra M, Schulz HH, Bakker J, van den Bemd BAT, van den Tol PM, Puijk RS, Lissenberg-Witte BI, de Gruijl TD, de Vries JJJ, Lagerwaard FJ, Scheffer HJ, Bruynzeel AME, Meijerink MR. MRI-guided stereotactic ablative body radiotherapy versus CT-guided percutaneous irreversible electroporation for locally advanced pancreatic cancer (CROSSFIRE): a single-centre, open-label, randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2024 May;9(5):448-459. doi: 10.1016/S2468-1253(24)00017-7. Epub 2024 Mar 19. PMID 38513683